CLINICAL TRIAL: NCT01137357
Title: Probiotics for Reduction Of Markers In Subjects With Allergy
Acronym: PROMISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Collaborators: Allergologiepraktijk Arnhem/Radboud/Rijnstate (Unknown); NIZO Food Research (Other); Wageningen University (Other); Campina Innovation (Unknown)
Responsible Party: Drs. A. Jansen, Allergologiepraktijk Arnhem/Radboud/Rijnstate
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTC 559-240908
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Hay Fever; Birch Pollen Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Yoghurt with Lactobacillus strain (L.plantarum WCFS1) (Experimental)
  Interventions: Dietary Supplement: Yoghurt with L. plantarum strain
- Yoghurt with Lactobacillus strain (L.plantarum NIZO3400) (Experimental)
  Interventions: Dietary Supplement: Yoghurt with L. plantarum strain
- Yoghurt with Lactobacillus strain (L. plantarum NIZO2877) (Experimental)
  Interventions: Dietary Supplement: Yoghurt with L. plantarum strain
- Yoghurt with Lactobacillus strain (L.plantarum CBS125632) (Experimental)
  Interventions: Dietary Supplement: Yoghurt with L. plantarum strain
- Yoghurt with Lactobacillus casei Shirota (Active Comparator)
  Interventions: Dietary Supplement: Yoghurt with L.casei
- Placebo Yoghurt (Placebo Comparator)
  Interventions: Dietary Supplement: Yoghurt

INTERVENTIONS:
Dietary Supplement: Yoghurt with L. plantarum strain — Intake of yoghurt during 4 weeks
  Arms: Yoghurt with Lactobacillus strain (L.plantarum WCFS1)
Dietary Supplement: Yoghurt with L.casei — Intake of yoghurt during 4 weeks
  Arms: Yoghurt with Lactobacillus casei Shirota
Dietary Supplement: Yoghurt with L. plantarum strain — Intake of yoghurt during 4 weeks
  Arms: Yoghurt with Lactobacillus strain (L.plantarum NIZO3400)
Dietary Supplement: Yoghurt with L. plantarum strain — Yoghurt with L. plantarum strain
  Arms: Yoghurt with Lactobacillus strain (L.plantarum CBS125632)
Dietary Supplement: Yoghurt with L. plantarum strain — Intake of yoghurt during 4 weeks
  Arms: Yoghurt with Lactobacillus strain (L. plantarum NIZO2877)
Dietary Supplement: Yoghurt — Intake of yoghurt during 4 weeks
  Arms: Placebo Yoghurt

SUMMARY:
In vitro studies reveal immunomodulatory effects of probiotic bacteria that are strain-dependent. Differential immunomodulatory in vitro capacities can not be extrapolated directly to in vivo efficacy. Thus, in vitro screening should be followed by comparative analysis of the selected immunomodulatory probiotic strains in an in vivo setting. Birch pollen allergy is one of the most common forms of respiratory allergy in European countries, and recognized by a Th2-skewed immune system. Five Lactobacillus strains will be evaluated for their immunomodulatory properties in birch pollen sensitive subjects outside the hay fever season. A double-blind placebo-controlled parallel study will be performed in which subjects with a proven birch pollen allergy will consume one of 5 different probiotic yoghurts containing 4 L. plantarum strains and 1 L. casei strain or a placebo yoghurt. Blood samples are collected at the start and after 4 weeks. Immune parameters are determined in serum and peripheral blood mononuclear cell cultures (hPBMC) derived from these subjects.

ELIGIBILITY:
Inclusion Criteria:

* birch pollen sensitive subjects
* Positive RAST or intracutane skintest
* age 18-50
* signed informed consent form

Exclusion Criteria:

* use of probiotics
* known allergy for pets (home setting)
* use of medication influencing the immune system
* use of antibiotics
* lactose intolerance
* pregnancy
* infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Il-13 in PBMC after ex-vivo stimulation with birch pollen allergen (Betv1)

SECONDARY OUTCOMES:
Other cytokines and cell-surface markers in PBMC ex vivo stimulation assay, birch pollen specific IgE, IgG and IgG4 in blood

CONTACTS AND LOCATIONS:
Overall Officials: A Jansen, Drs, Principal Investigator — Allergologiepraktijk Arnhem/Radboud/Rijnstate
Locations (1):
- Allergologiepraktijk Arnhem/Radboud/Rijnstate, Arnhem, Gelderland, Netherlands